CLINICAL TRIAL: NCT07087223
Title: The Open-Label, Multicenter Phase Ib/II Clinical Study Evaluating the Safety and Efficacy of Vebreltinib Combined With Furmonertinib in Locally Advanced or Metastatic NSCLC Patients With c-Met Amplification After EGFR-TKI Failure
Brief Title: Phase Ib/II Study of Vebreltinib With Furmonertinib in NSCLC Patients With c-Met Amplification After EGFR-TKI Failure
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024YJZ133
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer NSCLC
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- phase Ib Dose Escalation (Experimental)
  Interventions: Drug: Vebreltinib combined with Furmonertinib
- phase Ib Dose Expansion (Experimental)
  Interventions: Drug: Vebreltinib combined with Furmonertinib
- phase II (Experimental)
  Interventions: Drug: Vebreltinib combined with Furmonertinib

INTERVENTIONS:
Drug: Vebreltinib combined with Furmonertinib — Vebreltinib 100mg/1500mg/200mg oral twice daily combined with Furmonertinib 80mg oral once daily
  Arms: phase Ib Dose Escalation
Drug: Vebreltinib combined with Furmonertinib — Vebreltinib 100mg/1500mg/200mg oral twice daily combined with Furmonertinib 80mg oral once daily. Based on the safety data from the completed dose cohorts, the investigators will involve the selection of 1-2 dose cohorts for further study. Approximately 10 additional subjects will be enrolled in the selected dose expansion cohort to determine the recommended dose for Phase II clinical trials.
  Arms: phase Ib Dose Expansion
Drug: Vebreltinib combined with Furmonertinib — RP2D of Vebreltinib as determined during Phase Ib oral twice daily combined with Furmonertinib 80mg oral once daily
  Arms: phase II

SUMMARY:
The goal of phase Ib study was to evaluate efficacy and tolerability of the combination of vebreltinib and furmonertinib in patients with locally advanced or metastatic non-small cell lung cancer with c-met amplification after failure of EGFR-TKI treatment; to determine the maximum tolerated dose (MTD), and to evaluate the dose-limiting toxicity (DLT) and (recommended Phase 2 dose) RP2D of vebreltinib with furmonertinib.

The goal of phase II study was to evaluate efficacy [overall response rate (ORR), progression-free survival (PFS), and so on] of vebreltinib and furmonertinib in patients with locally advanced or metastatic non-small cell lung cancer with c-met amplification after failure of EGFR-TKI treatment.

DETAILED DESCRIPTION:
Phase Ib study uses 3+3 clinical design. The Phase Ib clinical trial is designed to explore the dosing of vebreltinib, consisting of two stages: dose escalation and dose expansion. The dose escalation stage follows a 3+3 design with three escalating dose levels (100 mg BID, 150 mg BID, 200 mg BID). Each dose cohort enrolls 3 patients. If no DLTs are observed in the first 3 patients within 28 days, the dose is escalated to the next cohort. If more than 1 DLT is observed in the first 3 patients within 28 days, that dose level is deemed non-tolerable. If 1 DLT is observed in the first 3 patients within 28 days, an additional 3 patients are enrolled at that dose level. If no DLTs are observed in the additional patients, dose escalation proceeds to the next cohort. If more than 1 DLT is observed among the additional patients (i.e., a total of 2 DLTs in the cohort), the previous dose level is determined to be the MTD. After completion of DLT assessment, the investigator decided whether to continue the treatment after the end of DLT assessment based on the subject 's tolerance and the safety profile of the dose group.

The dose expansion phase, based on the safety data from the completed dose cohorts, will involve the selection of 1-2 dose cohorts by the investigators for further study. Approximately 10 additional subjects will be enrolled in each selected dose expansion cohort to determine the recommended dose for Phase II clinical trials.

In the Phase II clinical study, the recommended Phase II dose of vebreltinib, determined from the Phase Ib study, will be combined with Furmonertinib to treat locally advanced or metastatic NSCLC with c-Met amplification in patients after failure of EGFR-TKI treatment. The study aims to evaluate the efficacy and safety of this combination, with an anticipated enrollment of 20 subjects. Participants will take vebreltinib (RP2D bid) and furmonertinib (80mg qd) until disease progression or undurable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Fully aware this study and voluntary to sign the informed consent form, and willing and able to comply with the study procedure.
2. Aged ≥18 years, male or female.
3. Patients with histologically or cytologically confirmed unresectable and non-suitable for radical surgery, or concurrent chemoradiotherapy , locally advanced or metastatic (stage IIIB, IIIC or IV) NSCLC;
4. Documented EGFR sensitive mutations (exon 19 deletion or exon 21 L858R mutation).
5. Disease progression after prior EGFR-TKI therapy. Participants must meet both of the following 2 criteria:

(1) ≤1 prior chemotherapy regimen allowed besides EGFR-TKI. Combination with anti-angiogenic therapy or PD-1/PD-L1 inhibitors are allowed during EGFR-TKI targeted therapy or chemotherapy.

（2） Objective clinical benefit documented during previous EGFR-TKI therapy, defined by either partial or complete radiological response, or durable stable disease should be greater than 6 months after initiation of EGFR-TKI.

6. After the last line of treatment before enrollment, progression is confirmed, and blood tests confirm c-Met amplification, or re-biopsy and genetic testing confirm c-Met amplification. Any of the following criteria define c-Met amplification.

1. For tumor tissue samples, FISH detection shows GCN ≥5 and/or MET/CEP7 ≥2 (FISH results from local testing institutions/central laboratories are acceptable);
2. Tissue (wax blocks from pleural effusion centrifugation, if quality-controlled) or blood NGS testing results confirm c-Met amplification with CN ≥2.3 (NGS results from local testing institutions/central laboratories are acceptable for both tissue and blood).

7. ECOG performance status ≤1. 8. According to RECIST v1.1, the patient must have at least one target lesion as assessed by the investigator.

9. Laboratory test results must meet the following criteria:

1. Absolute neutrophil count ≥1.5×10⁹/L (without the use of growth factors within 7 days prior to the start of treatment);
2. Hemoglobin ≥90 g/L (without blood transfusion or use of growth factors within 7 days prior to the start of treatment);
3. Platelet count ≥75×10⁹/L (without blood transfusion or use of growth factors within 7 days prior to the start of treatment);
4. Serum total bilirubin ≤1.5×upper limit of normal (ULN);
5. Serum alanine aminotransferase and aspartate aminotransferase ≤3×ULN (for patients with liver metastases, both AST and ALT ≤5×ULN);
6. Creatinine clearance (Ccr) ≥60 mL/min.
7. International normalized ratio (INR) ≤1.5×ULN;
8. Asymptomatic serum amylase ≤Grade 2 (NCI-CTCAE v5.0). For patients with Grade 2 serum amylase abnormalities at the start of the study, it must be confirmed that there are no signs and/or symptoms suggestive of pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal pancreatic imaging results);
9. Serum lipase ≤1.5×ULN. 10. Men with reproductive potential and women of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 3 months after the last dose of the study drug. Women of childbearing potential must have a negative serum pregnancy test within ≤7 days prior to the first dose of the study drug. This does not apply to female subjects who have undergone sterilization or are postmenopausal.

11. Expected survival ≥3 months.

Exclusion Criteria:

1. Patients with ALK fusion or ROS1 fusion.
2. Patients with spinal cord compression, leptomeningeal metastasis, or symptomatic brain metastasis that requires an increase in steroid dosage to control central nervous system disease. Patients with symptomatic CNS metastases that have been controlled may be eligible for this trial.
3. Presence of other malignancies (with the exception of any type of carcinoma in situ that has been completely resected, basal cell and squamous cell skin cancers, or other tumors/cancers that have been treated with curative intent and have been disease-free for at least 3 years).
4. A history of anti-tumor treatment that meets any of the following criteria:

（1）Received traditional Chinese medicine or patent medicine with anti-tumor indications within 1 week prior to the first dose of the study drug; （2）Underwent radiotherapy targeting the lung fields and whole brain within 4 weeks prior to the first dose of the study drug, or received radiotherapy targeting other areas (excluding the lung fields and whole brain) within 2 weeks prior to the first dose. Palliative radiotherapy for bone metastases to relieve pain or prevent skeletal-related events is excluded; （3）Underwent major surgery within 4 weeks, or has not recovered from the adverse effects of these surgeries. Thoracoscopic biopsy and mediastinoscopy are not considered major surgeries, and patients may be enrolled ≥1 week after the procedure 5. Has not recovered from any toxicity or complications of prior chemotherapy, surgery, radiotherapy, or other anti-tumor treatments, i.e., not reduced to ≤Grade 1 (NCI-CTCAE v5.0), with the exception of alopecia and permanent radiation-induced damage that cannot be recovered; 6. Requires the use of strong inhibitors or inducers of cytochrome P450 3A4 enzyme 1 week prior to the first dose of the study drug and during the study period.

7. Has any severe or uncontrolled systemic disease, including but not limited to:

1. Uncontrolled hypertension, with the allowance for the initiation or adjustment of antihypertensive medications prior to screening;
2. Positive for anti-HIV, or positive for both anti-HCV and HCV-RNA, or positive for HBsAg with HBV-DNA ≥500 IU/mL
3. Active keratitis or ulcerative keratitis during the disease phase;
4. Active tuberculosis;
5. Active infection requiring systemic antimicrobial therapy within 2 weeks prior to the first dose of the study drug;
6. Other severe medical conditions or psychiatric disorders, or laboratory abnormalities that, in the investigator's judgment, make the study drug unsuitable for the patient or affect protocol compliance; 8. Cardiac dysfunction and diseases that meet any of the following criteria:

（1）The average corrected QT interval calculated by the Fridericia formula from three electrocardiograms during the screening period >470 ms; （2）Any significant arrhythmias, such as ventricular arrhythmias, uncontrolled supraventricular or junctional arrhythmias, and other uncontrolled cardiac arrhythmias （3）Any risk factors for QTc prolongation, such as severe hypokalemia, hereditary long QT syndrome, or use of drugs that prolong the QT interval; d) Congestive heart failure with New York Heart Association (NYHA) classification ≥3; echocardiography indicating left ventricular ejection fraction (LVEF) <50%； 9. History of interstitial lung disease, drug-induced interstitial lung disease, or radiation pneumonitis requiring corticosteroid therapy, or is currently receiving drug therapy or other clinical interventions, or has active interstitial lung disease; 10. Has coagulation dysfunction or bleeding tendency 11. Has difficulty swallowing, or has active gastrointestinal disease, or has undergone major gastrointestinal surgery that may significantly affect the intake or absorption of the study drug 12. Has pleural effusion, pericardial effusion, or ascites that require drainage and/or are associated with dyspnea within 4 weeks prior to the first dose of the study drug; 13. Has any clinically significant systemic disease that requires treatment, as judged by the investigator, including but not limited to thyroid disease, organ transplant recipients, history of psychiatric disorders, history of drug abuse/addiction, alcoholism, or drug use; 14. History of acute or chronic pancreatitis, pancreatic surgery, or risk factors that may increase the risk of pancreatitis; 15. Patients receiving thrombolytic therapy are not eligible for inclusion, but patients receiving anticoagulant therapy may be included, provided that they have been on a stable dose of anticoagulant therapy for at least 1 week prior to the first dose; 16. Has a known hypersensitivity to the study drug or its excipients; 17. Pregnant or breastfeeding women; 18. Currently enrolled in another study device or study drug treatment, or received other study drugs or study devices within 2 weeks prior to the first dose of the study drug; 19. Cognitive impairment that may limit their understanding or execution of the informed consent form; 20. Presence of any condition that may increase the risk associated with the administration of the study drug, or may affect the interpretation of study results, or poor compliance with the study protocol, or any other situation that the investigator deems unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
phase Ib: Incidence of dose-limiting toxicities (DLT) as defined in the protocol | 12 months
  To determine the maximum tolerated dose (MTD) and/or dose-limiting toxicities (DLT) of combination therapy of Vebreltinib combined with Furmonertinib in locally advanced or metastatic NSCLC patients with c-Met amplification after EGFR-TKI failure
phase Ib: maximum tolerated dose (MTD) | 12 months
  To determine the maximum tolerated dose (MTD) and/or dose-limiting toxicities (DLT) of combination therapy of Vebreltinib combined with Furmonertinib in locally advanced or metastatic NSCLC patients with c-Met amplification after EGFR-TKI failure
phase Ib: Recommended Phase II Dose (RP2D) | 12 months
  To determine the recommended phase II dose (RP2D) of Vebreltinib in combination with Furmonertinib in locally advanced or metastatic NSCLC patients with c-Met amplification after EGFR-TKI failure
phase II: Overall Response Rate (ORR） | 24 months
  ORR is defined as the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1

SECONDARY OUTCOMES:
phase II: Progression Free Survival(PFS) | 24 months
  PFS is defined as the time from the first dose until the first documentation of progression or death from any cause, whichever occurs first, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
phase II: Duration of Response(DOR) | 24 months
  DOR is defined as the time from the first occurrence of a objective response to the time of documented disease progression, or death from any cause, whichever comes first, as assessed by the investigator using RECIST v1.1
phase II: Disease Control Rate(DCR) | 24 months
  DCR is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD), as assessed by the investigator using RECIST v1.1.
phase II: Overall Survival(OS) | 60 months
  OS is defined as the time from first dose until the date of death due to any cause
phase II: adverse events | Through study completion, an average of 2 year
  Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), etc, which includes laboratory tests, physical exams, electrocardiogram results and vital signs, according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
phase II: health-related quality of life | through study completion, an average of 2 year
  An EQ-5D-5L health survey questionnaire will be conducted before treatment, at each visit, and at the end of treatment to assess the impact of treatment on the patient's disease-related symptoms and health-related quality of life. The questionnaire will stop once the patient withdraws from the study. The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L profile defines health in terms of mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has five levels: 1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, and 5: extreme problems. The responses were used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 was the worst health you can imagine and 100 was the best health you can imagine.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Ordos Central Hospital, Neimeng, Neimeng
  - Peking University Cancer Hospital (Inner Mongolia Campus), Neimeng, Neimeng
  - Affiliated Hospital of Hebei University, Baoding
  - Baotou Cancer Hospital, Baotou
  - Peking University Cancer Hospital & Institute, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Beijing Daxing District People's Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Second Hospital of Dalian Medical University, Dalian
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No